CLINICAL TRIAL: NCT03351465
Title: A Randomized Controlled Trial of Coordinated Anxiety Learning and Management (CALM) for Pregnant and Postpartum Women
Brief Title: CALM for Pregnant and Post-Partum Women
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial was suspended due unanticipated funding issues.
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Christine Dunkel Schetter, PhD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CALM RCT
Record Dates: First submitted 2017-10-17; First posted 2017-11-22 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Anxiety; Depression; Depression, Postpartum; Pregnancy Related; CBT
MeSH Terms: conditions — Anxiety Disorders; Depression; Depression, Postpartum | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants will be recruited and randomized to the CALM intervention delivered in their homes or to treatment as usual.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CALM (Experimental): The intervention for this study, CALM Tools for Living-Il, is a computer-assisted cognitive-behavioral therapy for anxiety and depression that guides both the patient and CALM specialist. It is a reformulation of CALM Tools for Living that directly incorporates our previously optional modules for depression into the main program. The computerized/internet format is designed to retain the fidelity of CBT when delivered by novice clinicians. The program is intended to be delivered in 6 to 8 sessions, although flexibility is allowed. Participants in the intervention group will be visited by the calm specialist weekly between 6 and 8 times prenatally;postpartum visits will vary based on continuing assessment of symptoms.
  Interventions: Behavioral: Coordinated Anxiety Learning and Management
- Treatment as Usual (No Intervention): Participants will receive pre-natal care as usual, and will be visited at 4 time points by the graduate student researchers: baseline, 12 weeks post baseline, and 10 weeks postpartum.

INTERVENTIONS:
Behavioral: Coordinated Anxiety Learning and Management — The intervention for this study, CALM Tools for Living-Il, is a computer-assisted cognitive behavioral therapy for anxiety and depression that guides both the patient and CALM specialist. It is a reformulation of CALM Tools for Living42 that directly incorporates our previously optional modules for depression into the main program. The computerized internet format is designed to retain the fidelity of CBT when delivered by novice clinicians. The program is intended to be delivered in 6 to 8 sessions, although flexibility is allowed.
  Arms: CALM

SUMMARY:
Anxiety and depression is common along pregnant mothers and has been found to increase risk for negative outcomes in both mothers and infants. These risks can include low infant birth weight, negative mother-infant interactions, and delayed developmental outcomes. Evidenced-based interventions to support pregnant women experiencing symptoms of depression or anxiety are not well studied or widely available, particularly for low-income women of color. These women may not have access to the type of healthcare that would best support their needs and/or they may not be familiar with or trust clinicians who deliver mental health interventions. The current randomized-controlled trial (RCT) aims to address these gaps in the literature by testing the feasibility and efficacy of a doula-supported, computer-assisted delivery of a cognitive behavioral therapy (CBT) intervention designed to reduce pregnancy-related anxiety, depression, and prevent perinatal mood disorders. The 120 participants in the study (60 Black women and 60 Hispanic/Latina women) will be randomized to either receive the Coordinated Anxiety Learning and Management (CALM) intervention (n=60) or treatment as usual (n=60). Participants assigned to the intervention will complete 6-8 sessions of CALM with a language and ethnically/racially-matched doula who has been trained as a CALM specialist in order to increase participant comfort and reduce the stigma associated with mental health services. Women in both groups will complete assessments of their pregnancy-related anxiety, general anxiety, depressive symptoms, and satisfaction with treatment (CALM or treatment as usual) at baseline, 12-weeks post-baseline, and 10-weeks post-birth. It is hypothesized that women assigned to the CALM intervention will have significantly less anxiety and depressive symptoms post-treatment and post-partum compared to the women assigned to treatment as usual. The results of the current RCT will be used to test the efficacy of the CALM intervention for pregnant women or color and to inform efforts for potential future scalability.

DETAILED DESCRIPTION:
Setting and Sample Women will be recruited from six clinics in Alameda County that provide prenatal care. In clinic settings, women will be approached by a trained and culturally sensitive research graduate student researchers (GSRs) to determine their interest and eligibility for CALM participation based on inclusion and exclusion criteria. A standard screening form will be used.

Second, participants who remain eligible on the above criteria will be screened at the same time for pregnancy anxiety, depressive and anxiety symptoms using standardized screening instruments. Participants will be asked to complete the measures on a computer/tablet. Their responses will be scored and they will be informed via a phone call if they are eligible for the study. Those who score above population cutoffs for risk of disorders on The Overall Anxiety Severity and Impairment Scale (OASIS), Edinburgh Perinatal Depression Scale (EPDS), the Pregnancy-Specific Anxiety Scale (PSAS) and/or the Pregnancy-Related Anxiety Scale (PRAS) are eligible for the study. Cutoffs are as follows:

1. Pregnancy Specific Anxiety 4 items Scale (cut off 15 or higher)
2. Pregnancy-Related Anxiety Scale (cut off 30 or higher)

b) OASIS (cut off of 8 or greater for positive screen for anxiety symptoms) c) EPDS if not obtained as normal procedures in clinic at that time (cut off of 12 or greater for positive screen for depression)

Third, a home visit (or visit in their location of preference) is then arranged for participants who remain eligible for research staff to do the Mini International Neuropsychiatric Interview in order to exclude any women with history of bipolar, psychosis, current addiction or current suicidality. CALM web-based CBT is not recommended for individuals with severe mental illness (e.g. bipolar disorder and psychosis) who need additional services and will be given referrals. If not excluded on this basis research staff will consent women into the RCT study, conduct a baseline assessment, and randomized to treatment (CALM intervention) or control (Treatment as Usual) at the same home visit. Randomization will be programmed within the RedCap system after participants completed their baseline assessment. The computerized randomization schema will use blocked-randomization to ensure that too many participants are not assigned to the CALM intervention at once. Participants will be provided with remuneration at the end of the home visit, regardless of whether they are found eligible and/or consent to participate in the study.

CALM Intervention (Treatment) Each CALM-trained doula (referred to in study as "CALM specialist") will be assigned to a single participant for the entirety of their participation in the RCT. Study participants randomized to CALM will be visited weekly or biweekly in their home or location of preference by a CALM specialist between 6 and 8 times prenatally. Sessions may extend into postpartum if needed as determined by the CALM specialist in conjunction with their supervisor. Additional visits will vary based on continuing assessment of symptoms.

The CALM program is interactive, with individualized data entered session by session (e.g., symptom scales, homework completion, fear hierarchies, response to exercises in session), that is sometimes retrieved at later points throughout the program (e.g., fear hierarchies). The interactive data entry provides a tool for objectively monitoring progress throughout the program and a method for assessing symptom improvement from one visit to the next. In addition, video vignettes are embedded throughout to demonstrate a therapist and patient working together on a specific skill or component of treatment. To reinforce what was learned in session, printouts of the session material (including patient's individualized information that is entered) are given to participants at the completion of each session, providing them with an individualized workbook that cumulates as they progress through the program. Participants can also access the program through a patient portal to obtain more education, guidance and forms. Also, each module ends with an assessment section in which patients rate their understanding of the material and answer quiz questions, and clinicians rate the patient's proficiency in implementing the specific cognitive behavioral skill. This assessment information guides the participant and CALM specialist as to whether to repeat the module or not.

During the intervention, the CALM specialist will sit side by side with the patient as they both view the program on screen (see CALM Tools for Living Video, www.chammp.org). The program provides a structure to guide the content of each visit, thereby enhancing the integrity with which cognitive and behavioral strategies are presented and implemented in the hands of novice clinicians. The CALM specialist guides the participants to read or talk about material on the screen, following the general outline of module presentation described above. Participants can read the information and then talk with the CALM specialist about what was read, and/or or they can summarize the information that is presented on screen to the participant, and then help them apply the information to their own situation.

In addition, the program prompts CALM specialists to engage in specific tasks repeatedly throughout each module. These tasks include (1) stating the goals of each visit (2) entering participant data (e.g., number of homework practices completed) (3) choosing which links to select based on relevance to the participant's target problem (e.g., link for how to apply cognitive restructuring to social anxiety versus depression) (4) instruction in and demonstration of skills of breathing and cognitive restructuring (5) designing home work practices between visits (5) reviewing and problem solving home work practices and (6) summarizing the information from each section of the program. CALM Specialists will have portable printers to leave a copy of the homework for the participants in the CALM group, regardless of whether they have internet access to do it online.

The CALM specialist is trained in advance to use the program skillfully, so that they can direct participants to which sections of the computerized treatment are most relevant to them; inquire about and assess the patient's understanding of the material; summarize and rephrase sections of the text as necessary to provide clarification; assist in the application of CBT principles to the participants' idiosyncratic thoughts and behaviors; and reinforce in-session skills practice and between-session assignment practice. Also, CALM specialists may choose to skip some modules and advance to other modules based on the needs of a given participant. CALM specialists will meet weekly by phone with a licensed clinical psychologist (Co-I) for supervision and to ensure optimal care.

Study participants in the treatment group will also complete assessments at baseline, 12-week post-baseline, and 10-week postpartum follow-ups.

Treatment as Usual (Control) Currently, participants who screen high on any of the anxiety or depression measures are referred to behavioral and/or mental health services in Alameda County using a public health department (ACPHD) generated list of providers. For the purposes of this study, this procedure will remain the treatment as usual. Study participants not randomized to CALM will receive treatment as usual (TAU) and will complete baseline, 12-week post-baseline, and 10-week postpartum follow-up assessments only.

Measures Several measures in addition to the scores on the OASIS, EPDS, PSAS, and PRAS will be used to describe the sample, examine treatment effects, and to evaluate the participant satisfaction with the CALM program. First, a screening survey will be completed in the clinic (OASIS, EPDS, PSAS, and PRAS). Next participant assessments will be administered at baseline, 12 weeks post-baseline, and 10 weeks postpartum for all participants. The baseline assessment will be conducted in the home (or location of preference) as described above). The two follow-up assessments will either be completed online or over the phone with a GSR, depending on the participant's preference. Remuneration will be sent after completion of each assessment.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking
* Black or Hispanic/Latina women
* Over the age of 18
* Live or work in Oakland, CA.

CALM eligibility is based on two levels of screening. First, participants who score above clinical cutoffs on Overall Anxiety Severity and Impairment Scale (OASIS) or on the Edinburgh Perinatal Depression Scale (EPDS), or on the Pregnancy Stress and Anxiety Scale (PSAS) are eligible . A second screen using the Mini-Mental State Examination (MMSE) is required , as CALM and CBT are only effective in specific conditions and is not recommended for individuals with severe mental illness (e.g. bipolar disorder and psychosis) or cognitive impairment.

Exclusion Criteria:

* Multiple gestation
* Serving as birth surrogate
* Used reproductive technology

Women will also be excluded if they do not meet the above criteria (i.e., they do not exceed the clinical cutoffs) or if they have a history of bipolar disorder or psychosis (treated within the past year).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Pregnancy Related Anxiety (composite will be created with anxiety and depression measures) | at baseline, 12-weeks post-baseline, at 10 weeks postpartum
  14 item Pregnancy Stress and Anxiety Scale (PSAS) that measures pregnancy related stress and anxiety
Change in General Anxiety (composite will be created with anxiety and depression measures) | at baseline, 12-weeks post-baseline, at 10 weeks postpartum
  14 items from the Anxiety and Stress subscales of the Depression, Anxiety and Stress Scale (DASS)
Change in Depression (composite will be created with anxiety and depression measures) | at baseline, 12-weeks post-baseline, at 10 weeks postpartum
  10 items from the Edinburgh Postnatal Depression Scale (EPDS) that measures postnatal depressive symptoms

SECONDARY OUTCOMES:
Change in Functional Impairment | at baseline, 12-weeks post-baseline, and at 10 weeks postpartum
  5 item Sheehan Disability Scale (SDS) that measures functional impairment in school/ work, social, and family life (0-10 with higher scores indicating more impairment) and 2 items assessing number of days in one week participant felt were lost or unproductive due to symptoms of anxiety or depression (1-7).
Treatment Satisfaction | 12-weeks post-baseline
  5 item Client Satisfaction questionnaire that measures a participants' satisfaction with the treatment they've been delivered

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Francisco, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dunkel Schetter C. Psychological science on pregnancy: stress processes, biopsychosocial models, and emerging research issues. Annu Rev Psychol. 2011;62:531-58. doi: 10.1146/annurev.psych.031809.130727. PMID 21126184
- [Background] Huizink AC, Mulder EJ, Buitelaar JK. Prenatal stress and risk for psychopathology: specific effects or induction of general susceptibility? Psychol Bull. 2004 Jan;130(1):115-42. doi: 10.1037/0033-2909.130.1.115. PMID 14717652
- [Background] Dole N, Savitz DA, Hertz-Picciotto I, Siega-Riz AM, McMahon MJ, Buekens P. Maternal stress and preterm birth. Am J Epidemiol. 2003 Jan 1;157(1):14-24. doi: 10.1093/aje/kwf176. PMID 12505886
- [Background] Kramer MS, Lydon J, Seguin L, Goulet L, Kahn SR, McNamara H, Genest J, Dassa C, Chen MF, Sharma S, Meaney MJ, Thomson S, Van Uum S, Koren G, Dahhou M, Lamoureux J, Platt RW. Stress pathways to spontaneous preterm birth: the role of stressors, psychological distress, and stress hormones. Am J Epidemiol. 2009 Jun 1;169(11):1319-26. doi: 10.1093/aje/kwp061. Epub 2009 Apr 10. PMID 19363098
- [Background] Orr ST, Reiter JP, Blazer DG, James SA. Maternal prenatal pregnancy-related anxiety and spontaneous preterm birth in Baltimore, Maryland. Psychosom Med. 2007 Jul-Aug;69(6):566-70. doi: 10.1097/PSY.0b013e3180cac25d. Epub 2007 Jul 16. PMID 17636150
- [Background] Andersson L, Sundstrom-Poromaa I, Bixo M, Wulff M, Bondestam K, aStrom M. Point prevalence of psychiatric disorders during the second trimester of pregnancy: a population-based study. Am J Obstet Gynecol. 2003 Jul;189(1):148-54. doi: 10.1067/mob.2003.336. PMID 12861154
- [Background] Ross LE, McLean LM. Anxiety disorders during pregnancy and the postpartum period: A systematic review. J Clin Psychiatry. 2006 Aug;67(8):1285-98. doi: 10.4088/jcp.v67n0818. PMID 16965210
- [Background] Lee AM, Lam SK, Sze Mun Lau SM, Chong CS, Chui HW, Fong DY. Prevalence, course, and risk factors for antenatal anxiety and depression. Obstet Gynecol. 2007 Nov;110(5):1102-12. doi: 10.1097/01.AOG.0000287065.59491.70. PMID 17978126
- [Background] Teixeira C, Figueiredo B, Conde A, Pacheco A, Costa R. Anxiety and depression during pregnancy in women and men. J Affect Disord. 2009 Dec;119(1-3):142-8. doi: 10.1016/j.jad.2009.03.005. Epub 2009 Apr 5. PMID 19346001
- [Background] Woods SM, Melville JL, Guo Y, Fan MY, Gavin A. Psychosocial stress during pregnancy. Am J Obstet Gynecol. 2010 Jan;202(1):61.e1-7. doi: 10.1016/j.ajog.2009.07.041. Epub 2009 Sep 20. PMID 19766975
- [Background] Gavin NI, Gaynes BN, Lohr KN, Meltzer-Brody S, Gartlehner G, Swinson T. Perinatal depression: a systematic review of prevalence and incidence. Obstet Gynecol. 2005 Nov;106(5 Pt 1):1071-83. doi: 10.1097/01.AOG.0000183597.31630.db. PMID 16260528
- [Background] Goodman SH. Depression in mothers. Annu Rev Clin Psychol. 2007;3:107-35. doi: 10.1146/annurev.clinpsy.3.022806.091401. PMID 17716050
- [Background] Bener A, Gerber LM, Sheikh J. Prevalence of psychiatric disorders and associated risk factors in women during their postpartum period: a major public health problem and global comparison. Int J Womens Health. 2012;4:191-200. doi: 10.2147/IJWH.S29380. Epub 2012 May 10. PMID 22654524
- [Background] Matthey S, Barnett B, Howie P, Kavanagh DJ. Diagnosing postpartum depression in mothers and fathers: whatever happened to anxiety? J Affect Disord. 2003 Apr;74(2):139-47. doi: 10.1016/s0165-0327(02)00012-5. PMID 12706515
- [Background] Yelland J, Sutherland G, Brown SJ. Postpartum anxiety, depression and social health: findings from a population-based survey of Australian women. BMC Public Health. 2010 Dec 20;10:771. doi: 10.1186/1471-2458-10-771. PMID 21167078
- [Background] Murray L, de Rosnay M, Pearson J, Bergeron C, Schofield E, Royal-Lawson M, Cooper PJ. Intergenerational transmission of social anxiety: the role of social referencing processes in infancy. Child Dev. 2008 Jul-Aug;79(4):1049-64. doi: 10.1111/j.1467-8624.2008.01175.x. PMID 18717906
- [Background] Stein A, Craske MG, Lehtonen A, Harvey A, Savage-McGlynn E, Davies B, Goodwin J, Murray L, Cortina-Borja M, Counsell N. Maternal cognitions and mother-infant interaction in postnatal depression and generalized anxiety disorder. J Abnorm Psychol. 2012 Nov;121(4):795-809. doi: 10.1037/a0026847. Epub 2012 Jan 30. PMID 22288906
- [Background] Dunkel Schetter C, Tanner L. Anxiety, depression and stress in pregnancy: implications for mothers, children, research, and practice. Curr Opin Psychiatry. 2012 Mar;25(2):141-8. doi: 10.1097/YCO.0b013e3283503680. PMID 22262028
- [Background] Lu Q, Lu MC, Schetter CD. Learning from success and failure in psychosocial intervention: an evaluation of low birth weight prevention trials. J Health Psychol. 2005 Mar;10(2):185-95. doi: 10.1177/1359105305049763. PMID 15723889
- [Background] Stevens-Simon C, Orleans M. Low-birthweight prevention programs: the enigma of failure. Birth. 1999 Sep;26(3):184-91. doi: 10.1046/j.1523-536x.1999.00184.x. PMID 10655819
- [Background] Butler AC, Chapman JE, Forman EM, Beck AT. The empirical status of cognitive-behavioral therapy: a review of meta-analyses. Clin Psychol Rev. 2006 Jan;26(1):17-31. doi: 10.1016/j.cpr.2005.07.003. Epub 2005 Sep 30. PMID 16199119
- [Background] Tolin DF. Is cognitive-behavioral therapy more effective than other therapies? A meta-analytic review. Clin Psychol Rev. 2010 Aug;30(6):710-20. doi: 10.1016/j.cpr.2010.05.003. Epub 2010 May 25. PMID 20547435
- [Background] Hodnett ED, Fredericks S, Weston J. Support during pregnancy for women at increased risk of low birthweight babies. Cochrane Database Syst Rev. 2010 Jun 16;(6):CD000198. doi: 10.1002/14651858.CD000198.pub2. PMID 20556746
- [Background] Sockol LE, Epperson CN, Barber JP. A meta-analysis of treatments for perinatal depression. Clin Psychol Rev. 2011 Jul;31(5):839-49. doi: 10.1016/j.cpr.2011.03.009. Epub 2011 Mar 27. PMID 21545782
- [Background] O'Mahen H, Himle JA, Fedock G, Henshaw E, Flynn H. A pilot randomized controlled trial of cognitive behavioral therapy for perinatal depression adapted for women with low incomes. Depress Anxiety. 2013 Jul;30(7):679-87. doi: 10.1002/da.22050. Epub 2013 Jan 14. PMID 23319454
- [Background] Andrews G, Cuijpers P, Craske MG, McEvoy P, Titov N. Computer therapy for the anxiety and depressive disorders is effective, acceptable and practical health care: a meta-analysis. PLoS One. 2010 Oct 13;5(10):e13196. doi: 10.1371/journal.pone.0013196. PMID 20967242
- [Background] Craske MG, Rose RD, Lang A, Welch SS, Campbell-Sills L, Sullivan G, Sherbourne C, Bystritsky A, Stein MB, Roy-Byrne PP. Computer-assisted delivery of cognitive behavioral therapy for anxiety disorders in primary-care settings. Depress Anxiety. 2009;26(3):235-42. doi: 10.1002/da.20542. PMID 19212970
- [Background] Roy-Byrne P, Craske MG, Sullivan G, Rose RD, Edlund MJ, Lang AJ, Bystritsky A, Welch SS, Chavira DA, Golinelli D, Campbell-Sills L, Sherbourne CD, Stein MB. Delivery of evidence-based treatment for multiple anxiety disorders in primary care: a randomized controlled trial. JAMA. 2010 May 19;303(19):1921-8. doi: 10.1001/jama.2010.608. PMID 20483968
- [Background] Craske MG, Stein MB, Sullivan G, Sherbourne C, Bystritsky A, Rose RD, Lang AJ, Welch S, Campbell-Sills L, Golinelli D, Roy-Byrne P. Disorder-specific impact of coordinated anxiety learning and management treatment for anxiety disorders in primary care. Arch Gen Psychiatry. 2011 Apr;68(4):378-88. doi: 10.1001/archgenpsychiatry.2011.25. PMID 21464362
- [Background] Sullivan G, Sherbourne C, Chavira DA, Craske MG, Gollineli D, Han X, Rose RD, Bystritsky A, Stein MB, Roy-Byrne P. Does a quality improvement intervention for anxiety result in differential outcomes for lower-income patients? Am J Psychiatry. 2013 Feb;170(2):218-25. doi: 10.1176/appi.ajp.2012.12030375. PMID 23377641
- [Background] Joesch JM, Sherbourne CD, Sullivan G, Stein MB, Craske MG, Roy-Byrne P. Incremental benefits and cost of coordinated anxiety learning and management for anxiety treatment in primary care. Psychol Med. 2012 Sep;42(9):1937-48. doi: 10.1017/S0033291711002893. Epub 2011 Dec 13. PMID 22152230
- [Background] Stanley D, Sata N, Oparah JC, McLemore MR. Evaluation of the East Bay Community Birth Support Project, a Community-Based Program to Decrease Recidivism in Previously Incarcerated Women. J Obstet Gynecol Neonatal Nurs. 2015 Nov-Dec;44(6):743-50. doi: 10.1111/1552-6909.12760. Epub 2015 Oct 15. PMID 26469292
- [Background] Hodnett ED, Gates S, Hofmeyr GJ, Sakala C, Weston J. Continuous support for women during childbirth. Cochrane Database Syst Rev. 2011 Feb 16;(2):CD003766. doi: 10.1002/14651858.CD003766.pub3. PMID 21328263
- [Background] Kozhimannil KB, Hardeman RR, Attanasio LB, Blauer-Peterson C, O'Brien M. Doula care, birth outcomes, and costs among Medicaid beneficiaries. Am J Public Health. 2013 Apr;103(4):e113-21. doi: 10.2105/AJPH.2012.301201. Epub 2013 Feb 14. PMID 23409910
- [Background] Rose RD, Lang AJ, Welch SS, Campbell-Sills L, Chavira DA, Sullivan G, Sherbourne C, Bystritsky A, Stein MB, Roy-Byrne PP, Craske MG. Training primary care staff to deliver a computer-assisted cognitive-behavioral therapy program for anxiety disorders. Gen Hosp Psychiatry. 2011 Jul-Aug;33(4):336-42. doi: 10.1016/j.genhosppsych.2011.04.011. Epub 2011 Jun 8. PMID 21762829
- [Background] Brown LA, Craske MG, Glenn DE, Stein MB, Sullivan G, Sherbourne C, Bystritsky A, Welch SS, Campbell-Sills L, Lang A, Roy-Byrne P, Rose RD. CBT competence in novice therapists improves anxiety outcomes. Depress Anxiety. 2013 Feb;30(2):97-115. doi: 10.1002/da.22027. Epub 2012 Dec 5. PMID 23225338